CLINICAL TRIAL: NCT05462223
Title: A Study of the Safety and Feasibility of the Vessel Restoration System for AVF to Promote the Physiologic and Functional Maturation of Upper-extremity Autologous End-to-Side Arteriovenous Fistulas (AVF) in Patients With Chronic Kidney Disease: ACTIVATE AVF
Brief Title: Alucent Vessel Restoration System for AVF
Acronym: Activate AVF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Alucent Biomedical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 1061-003
Record Dates: First submitted 2022-07-08; First posted 2022-07-18 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: AV Fistula
MeSH Terms: conditions — Arteriovenous Fistula

STUDY DESIGN:
Intervention Model Description: A prospective, single-arm, multicenter, open-label study of the VRS-AVF for use as adjunctive therapy in the surgical creation of an end-to-side brachiocephalic (BC) AVF.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Alucent VRS for Treatment of Atherosclerotic Lesions (Experimental): Alucent Vessel Restoration System for AVF (VRS-AVF) consists of the following components:
  1. VRS 10-8-10 Dimer Coated Balloon Catheter for AVF
  2. VRS Light Fiber
  3. VRS Light Source
  Interventions: Combination Product: Alucent Vessel Restoration System for AVF

INTERVENTIONS:
Combination Product: Alucent Vessel Restoration System for AVF — Alucent Vessel Restoration System for AVF (VRS-AVF) consists of the following components:
  1. VRS 10-8-10 Dimer Coated Balloon Catheter for AVF
  2. VRS Light Fiber
  3. VRS Light Source

SUMMARY:
Feasibility of the Vessel Restoration System for AVF

DETAILED DESCRIPTION:
A study of the safety and feasibility of the Vessel Restoration System for AVF to promote the physiologic and functional maturation of a Brachiocephalic End-to-Side Arteriovenous Fistulas (AVF) in Patients with Chronic Kidney Disease Stage V (Pre-dialysis): ACTIVATE AVF

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and can provide informed consent
* Use birth control
* Chronic Kidney Disease

Exclusion Criteria:

* Receiving hemodialysis
* Pregnant, breastfeeding, planning to become pregnant
* Receiving immunosuppressants
* Has "Long COVID"

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-07-15 (Actual); Primary Completion 2024-05-15 (Estimated); Study Completion 2024-12-15 (Estimated)

PRIMARY OUTCOMES:
AVF Maturation | 2 weeks to 3 months
  Unassisted AVF Maturation using a fistulagram and needle sticks to assess maturation at specific time points

CONTACTS AND LOCATIONS:
Locations (12):
- Australia (8):
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Prince of Wales, Randwick, New South Wales
  - Royal North Shore Hospital & North Shore Private, Saint Leonards, New South Wales
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Flinders Medical Center, Bedford Park, South Australia
  - The Alfred Hospital, Melbourne, Victoria
  - Northern Health, Richmond, Victoria
  - Royal Perth Hospital, Perth, Western Australia
- Poland (4):
  - Poznan University of Medical Sciences, Lublin
  - Wojskowy Instytut Medczny z Centrainym Szpitalem Klinicznym Ministerstwa Obrony Narodowej, Warsaw
  - Lower Silesia Center of Heart Diseases MEDINet, Wroclaw
  - Klincznny Oddzial Chirurgii Naczyniowej Szpital Uniweryzstecki w Zielonej, Zielona Góra